CLINICAL TRIAL: NCT00137293
Title: A Study to Characterize the Acute Electrophysiologic Properties, Safety and Tolerability of GAP-486
Brief Title: Study Evaluating GAP-486 in Heart Rhythm
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 3163K1-201
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Arrhythmia
Keywords: Arrhythmia, syncope, antiarrhythmic
MeSH Terms: conditions — Arrhythmias, Cardiac; Syncope | interventions — rotigaptide; Sodium Chloride

INTERVENTIONS:
Drug: GAP-486 (ZP-123)
Drug: 0.9% Sodium Chloride, USP

SUMMARY:
The purpose of this study is to learn the effects of a test drug on heart rhythm, and to provide additional data to see if the test drug is well tolerated and safe.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an electrophysiology study for evaluation of heart rhythm.

Exclusion Criteria:

* Patients with uncontrolled blood pressure
* Patients with certain cardiac risk factors
* Patients with significant kidney or liver problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-11; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
This study takes place within 24 hours. The measure to determine the effect of the intervention will be the difference in values from the baseline electrophysiology study, and the values obtained after intervention within the test drug.

SECONDARY OUTCOMES:
This study takes place within 24 hours, and looks at the changes in values of electrophysiology studies, before and after administration of test article.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (6):
- United States (3):
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Hershey, Pennsylvania
- Canada (3):
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec